CLINICAL TRIAL: NCT03829735
Title: Neonatal Vaccination Against Hepatitis B in Africa - Sero-survey in Senegal
Acronym: NeoVac2S
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not started
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-048
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children and their mothers (Experimental): Human biological samples from children aged 9 to 12 months and their mothers. Capillary and venous blood samples.
  Interventions: Other: Human biological samples

INTERVENTIONS:
Other: Human biological samples — Collection of capillary blood for HbsAg testing. Collection of 12 mL of blood for HbsAg positive women and 1 mL for HbsAg positive children.

SUMMARY:
Chronic infection with hepatitis B virus (HBV) is a leading cause of death in adults in sub-Saharan Africa (SSA). Prior to the introduction of the hepatitis B vaccine, main modes of transmission in SSA were perinatal transmission from mother-to-child (MTCT) (10%) and horizontal transmission during early childhood (90%). MTCT occurs through contact with maternal fluids during passage through the birth cana; transplacental transmission and transmission through breastfeeding are rare.

In 2009, WHO recommended the administration of hepatitis B vaccination to all newborns within 24 hours of birth to prevent perinatal and early transmissions. In Senegal, the government introduced the monovalent vaccine that can be used within 24 hours after birth in the Expanded Program on Immunization (EPI) in March 2016.

Here, we present a study protocol for a sero-epidemiological study of pairs of children aged 9 to 12 months and their mothers, identified through the demographic study, to assess the impact of monovalent vaccine introduced by the national program for prevention of mother-to-child transmission in Senegal. We will also assess the diagnostic performance of loop-mediated isothermal amplification assay (LAMP) to identify people with high viral replication (HBV DNA ≥200,000 IU/ml), compared to a conventional reference test (PCR).

DETAILED DESCRIPTION:
Chronic infection with hepatitis B virus (HBV) is a leading cause of death in adults in sub-Saharan Africa (SSA). Each year, about 61,000 people are estimated to die of hepatocellular carcinoma (HCC) or cirrhosis secondary to chronic infection with HBV. Prior to the introduction of the hepatitis B vaccine, main modes of transmission in SSA were perinatal transmission from mother-to-child (MTCT) (10%) and horizontal transmission during early childhood (90%). MTCT occurs through contact with maternal fluids during passage through the birth cana; transplacental transmission and transmission through breastfeeding are rare.

Despite a relatively low frequency of perinatal transmission in SSA, prevention of this type of transmission is important, because this mode of transmission results in higher risk of becoming chronic HBV carriers, and developing chronic liver disease, including HCC, than horizontal transmission.

In 2009, WHO recommended the administration of hepatitis B vaccination to all newborns within 24 hours of birth to prevent perinatal and early transmissions. In Senegal, the government introduced the monovalent vaccine that can be used within 24 hours after birth in the Expanded Program on Immunization (EPI) in March 2016.

It is in this context that the NeoVac study started in 2016 in Senegal, Burkina Faso and Madagascar. The general objective is to develop a long-term strategy adapted to the local context to vaccinate newborns against hepatitis B in the first 24 hours of life.

The NeoVac 1, a population-based epidemiological survey to estimate the coverage of this newly introduced monovalent hepatitis B vaccine started in Senegal in 2018. Here, we present a study protocol for a sero-epidemiological study of pairs of children aged 9 to 12 months and their mothers, identified through the demographic study, to assess the impact of monovalent vaccine introduced by the national program for prevention of mother-to-child transmission in Senegal. We will also assess the diagnostic performance of loop-mediated isothermal amplification assay (LAMP) to identify people with high viral replication (HBV DNA ≥200,000 IU/ml), compared to a conventional reference test (PCR).

ELIGIBILITY:
Inclusion Criteria:

All mothers of children between 9 and 12 months of age registered in the SSDS of Niakhar, Bambey and Fatick, who accept a blood sample from her and their child.

Exclusion Criteria:

* A child without a mother identified for sampling
* Failure to sign informed consent to participate in the NeoVac 2 study

Min Age: 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Vaccination coverage of the vaccine at birth from the health record and health post registers | 9 to 12 months post-natal visit
  Collection of thedate of vaccination of children aged 9-12 months

SECONDARY OUTCOMES:
Positive HBsAg among mothers of children aged 9-12 months | 9 to 12 months post-natal visit
  HBsAg testing from capillary blood on site
Positive HBsAg among children aged 9-12 months | 9 to 12 months post-natal visit
  HBsAg testing from capillary blood on site

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Taieb, Principal Investigator — Institut Pasteur Dakar

IPD SHARING:
Plan to Share IPD: No